CLINICAL TRIAL: NCT07242352
Title: Dynamic Marker - Adjusted Therapy Comparing Adjuvant Elacestrant With Standard Endocrine Treatment in Genomically and/or Clinically High-risk ER+/HER2- Early Breast Cancer (ADAPTela)
Brief Title: Marker - Adjusted Therapy Comparing Adjuvant Elacestrant With Standard Endocrine Treatment in Genomically and/or Clinically High-risk ER+/HER2- eBC
Acronym: ADAPTela
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Berlin-Chemie Menarini (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM16 (ADAPTela); 2025-522484-15-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; HR+/HER2- Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant

STUDY DESIGN:
Intervention Model Description: This is a multicentre, interventional, prospective, two-arm, randomised, open-label, controlled adjuvant, phase III-trial evaluating the efficacy and safety of elacestrant (combined with ribociclib, if applicable) versus standard-of-care (SoC) endocrine therapy (ET) in HR+/HER2- early breast cancer (eBC) patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elacestrant upfront (ELA) (Experimental): Patients will be treated with elacestrant (ELA) for 5 years. In case further treatment, e.g., CDK4/6 inhibitors, is indicated, ribociclib (RIBO) may be added for 3 years in parallel
  Interventions: Drug: Elacestrant
- Standard-of-care endocrine treatment (SoC-ET) (Active Comparator): Patients will be treated with SoC ET for 5-10 years. In case further treatment, e.g., CDK4/6 inhibitors, is indicated, this may be added according to SoC and per investigator´s discretion.
  Interventions: Drug: Standard-of-care endocrine treatment

INTERVENTIONS:
Drug: Elacestrant — Elacestrant, a tetrahydronaphthalene compound, is a potent, selective, and orally active oestrogen receptor-α (ERα) antagonist and degrader.
  Other Names: ORSERDU
  Arms: Elacestrant upfront (ELA)
Drug: Standard-of-care endocrine treatment — SoC ET comprises all endocrine treatments authorized for the condition under review. The choice is made upon investigator´s discretion.
  Arms: Standard-of-care endocrine treatment (SoC-ET)

SUMMARY:
In this clinical trial, the Sponsor plans to investigate whether patients with HR+/HER2- eBC identified during routine clinical assessments and treatments as having intermediate to high-risk (based on Oncotype DX® or similar tests and on response assessment to 2-6 weeks of preoperative ET) achieve a survival benefit from an initial 5-years use of elacestrant (with or without a CDK 4/6 inhibitor) followed by SoC ET for further 0-2.5 years in comparison to at least 5 up to 7.5 years SoC ET therapy (+/- CDK4/6 inhibitor).

Based on several studies in the metastatic setting, it is reasonable to assume that the adjuvant use of elacestrant with or without CDK 4/6 inhibitors will prevent or delay the activation of mechanisms conferring resistance to ET (e.g., ESR1 mutations).

DETAILED DESCRIPTION:
Patients with hormone-receptor positive/HER2-negative (HR+/HER2-) early breast cancer (eBC) remain at risk of recurrence for many years after diagnosis. Current guidelines provide treatment recommendations depending on stage, histological grade, and menopausal status. However, patients with a high-risk HR+/HER2- eBC are at need for more efficacious treatment.

Several new strategies are currently investigated in patients diagnosed with high-risk HR+/HER2- eBC, including extending the duration of adjuvant endocrine therapy (ET), addition of ovarian function suppression (OFS) in case of premenopausal patients, and intensification of adjuvant ET by use of new therapies, such as cyclin-dependent kinase (CDK) 4/6 inhibitors. Moreover, development of algorithms incorporating not only clinical variables, but also key tumor biological variables such as Oncotype DX®/Recurrence Score (RS) or Mammaprint®, and possibly dynamic variables such as ET-response measured by Ki-67 after 2-6 weeks of preoperative standard endocrine induction therapy, could be of immense importance for risk estimation and subsequently optimization of therapy in intermediate to high-risk patients.

Several retrospective studies have shown that Oncotype DX® or other genomic tests are informative regarding prediction of treatment benefit in HR+/HER2- eBC. Therefore, use of RS instead of mostly relying on histological grade provides stronger prognostic and predictive information.

Further, characterization of ET-response has shown to provide important prognostic information in early HR+/HER2- eBC beyond clinical and genomic markers, as shown in the WSG-ADAPT-HR+/HER2-, ALLIANCE, and POETIC trials. The endocrine response has therefore become part of the ESMO guidelines as a prognostic factor.

The combination of classical prognostic markers with genomic assessments (e.g., Oncotype DX®) and endocrine response seems to be the most promising tool for identification of patients with significant relapse risk despite of standard ET and/or chemotherapy.

Remarkably in the 5-year analysis of the WSG-ADAPT-HR+/HER2- trial, ET-responders with RS >25 were shown to have more favorable survival than ET-non-responders, despite of higher pCR-rates in a subset of neoadjuvant chemotherapy (NACT)-treated patients. Therefore, patients with high genomic or clinical risk and/or ET-non responders with RS >25 with intermediate clinical risk are at need for alternative, more efficacious treatment approaches.

Optimal ET treatment in patients with intermediate-risk stage I-II disease but enhanced relapse risk remains unclear despite of the significant positive impact of Ribociclib on iDFS in stage II-patients demonstrated in NATALEE (NCT03701334).

The ADAPTcycle trial, based on the positive results for CDK 4/6 inhibitors in the adjuvant setting as shown in the MonarchE and NATALEE trials [12], is currently investigating whether replacing chemotherapy by an ET-CDK 4/6 based approach could be a better option for particular subgroups which are identified by combination of clinical and genomic risk and ET-responder status.

Moreover, the ongoing ADAPTlate trial investigates the impact of abemaciclib if added to standard ET in intermediate to high-risk HR+/HER2- eBC given immediately or within the first 2-6 years after completion of primary therapy.

Elacestrant is a novel, nonsteroidal, oral, selective oestrogen receptor degrader (SERD) that inhibits oestradiol-dependent gene transcription downstream of ER, including its mutated receptor variants, which is associated with endocrine resistance as demonstrated in phase I-trials [13]. Therefore, adjuvant use of SERDs may be beneficial in preventing ET resistance mechanisms.

In the phase III-trial EMERALD (NCT03778931), elacestrant improved PFS vs SoC in patients with metastatic HR+/HER2- breast cancer previously treated with ET in combination with a CDK4/6 inhibitor, especially in those harboring an ESR1-mutation. Also, according to EMBER-3 data in the metastatic setting, the use of SERDs in combination with standard CDK 4/6 inhibitors in patients with stage II-disease may be particularly effective across mutational profiles.

Interestingly, other SERDs were shown to yield a PFS benefit specificity in subgroups with mutated ESR1 variants and appear to require a combination with CDK 4/6 inhibitors to improve survival in wild-type ESR1 receptors, as demonstrated in the EMBER-3 trial.

Elacestrant is also under investigation in eBC. The phase I trial ELIPSE (NCT04797728) in postmenopausal women with early-stage (stage cT1-3, N0), ER-positive, HER2-negative breast cancer investigates 400 mg of elacestrant daily for four weeks in the neoadjuvant setting. The trial's primary outcome is proliferation arrest, defined as a Ki-67 level of ≤ 2.7%, in the surgical specimens collected after the end of trial treatment. Furthermore, the EORTC-2129-BCG (TREAT ctDNA, NCT05512364) is a phase III trial in pre- and postmenopausal women and men with high-risk early-stage ER-positive, HER2-negative breast cancer, and circulating tumor DNA (ctDNA) relapse. ctDNA-positive patients identified during the eligibility assessment, with no evidence of distant metastasis, will be randomized to receive either SoC endocrine treatment or elacestrant; the trial's primary endpoint is distant metastasis-free survival. However, this trial focuses on the populations at a high risk of recurrence, that is, stage IIB or stage III disease and completion of adjuvant chemotherapy or patients with at least four cycles of neoadjuvant chemotherapy and residual tumor at surgery of ≥ 1cm (≥ypT1c) or axillary node-positive (ypN+). Therefore, the information provided by the EORTC-2129-BCG trial on the activity of elacestrant in patients with intermediate-risk stage I-II disease will be limited.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, independent from gender
2. Patient must be ≥18 years at diagnosis
3. The patient must be capable of giving informed consent and be willing and able to comply with the requirements and restrictions in this protocol and accessible for treatment and follow-up
4. Sign informed consent prior to any study-specific procedures.
5. Histologically confirmed unilateral, primary invasive carcinoma of the breast Note: bilateral, multicentric, or multifocal carcinoma may only be included after consultation of Sponsor.
6. Histologically confirmed diagnosis of primary hormone-receptor-positive (HR+) (i.e., oestrogen-receptor (ER) ≥ 10% and progesterone-receptor PR ≥ 10%) early breast cancer by local laboratory Note: ER positive according to ASCO / AGO Guidelines, ER 1-10% (low) is not defined as HR+.
7. Patient has HER2-negative breast cancer defined as a negative in-situ hybridization test or an IHC status of 0, 1+, or 2+, if IHC is 2+, a negative in-situ hybridization (FISH, CISH, or SISH) test is required (based on the most recently analysed tissue sample and all tested by a local laboratory).
8. No evidence of distant metastasis (confirmed by CT thorax / abdomen, X-ray chest, ultrasound liver, bone scan, or PET-CT, respectively, performed within clinical routine).
9. High genomic risk assessment within clinical routine (Oncotype DX® preferred; In those cases, where Oncotype Dx® is not possible in clinical routine, Oncotype Dx® should be assessed retrospectively after inclusion of the patient and as a study specific measure, provided sufficient tumour tissue from primary diagnosis is available.)
10. 10. Completed 2-6 weeks of endocrine induction treatment and Ki-67 response assessment Note: 2-4 weeks recommended, up to 6 weeks allowed. Endocrine induction is highly recommended, but if endocrine induction therapy could not be performed or ET response is not representative, clinical factors should be used.
11. 11. Completed (neo)adjuvant chemotherapy, if applicable
12. Completed radiotherapy, if applicable
13. Patient meets any of the following three conditions at end of primary treatment (including endocrine induction treatment, biopsy/surgery, and if necessary, chemotherapy and radiotherapy and up to 12 months standard-of-care endocrine treatment, excluding previous treatment > 4 weeks with any SERD):

    Pathological Stage * Genomical High-Risk (Oncotype Dx®)** Age Clinical High-Risk Factors Stage I T1 N0

    RS>25 Any age High risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * No Chemotherapy
    * G3 or PR negative and Ki-67 >25%***
    * Non-pCR after NACT*

    RS 16-25 Age <50 High risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * No Chemotherapy
    * G3 or PR negative and Ki-67 >25%***
    * Non-pCR after NACT* Any genomic risk Any age G3 and Ki-67>40%

    Stage IIa with T2 N0

    RS 0-25 Age>50 High risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * G3 and Ki-67>40%
    * G3 or PR negative and Ki-67 >25%***
    * Non-pCR after NACT*

    RS 0-15 Age<50 No chemotherapy AND high risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * G3 and Ki-67>40%
    * G3 or PR negative and Ki-67 >25%***
    * Non-pCR after NACT*

    RS 16-25 Age<50 No chemotherapy, AND/OR high risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * G3 and Ki-67>40%
    * G3 or PR negative and Ki-67 >25%***
    * Non-pCR after NACT*

    RS >25 Any age Any clinical risk

    Any genomic risk Any age G3 and Ki-67 >40%

    Stage IIa with T1 N1, G1-2

    RS 0-25 Age>50 High risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * PR negative and Ki-67 >25%***
    * Non-pCR after NACT*
    * 3 positive LN

    RS 0-25 Age <50 No chemotherapy, AND/OR high risk (≤ 1 factor applies):
    * ET non-response (post ET Ki-67 >10%)***
    * PR negative and Ki-67 >25%***
    * Non-pCR after NACT*
    * 3 positive LN

    RS>25 Any age Any clinical risk

    Stage IIb with T3 N0 or T2 N1, G1-2 Any genomic risk Any age Any clinical risk

    * In patients treated by neoadjuvant chemotherapy, clinical stage should be used for inclusion

    ** In stage I-IIa and N0 patients with unknown genomic risk prior to inclusion, Oncotype Dx® Test should be performed on untreated tumour tissue within clinical routine.

    Results of other genomic tests, if already performed within the clinical routine, may be considered. In such cases, inclusion is only possible if clinical high-risk criteria apply and after consultation with sponsor.

    In those cases, where Oncotype Dx® is missing from clinical routine and in the N1-situation, Oncotype Dx® should be assessed retrospectively after inclusion of the patient and as a study specific measure, provided sufficient tumour tissue from primary diagnosis is available.

    *** Use of clinical factors is recommended in patients with unknown or not representative ET response.
14. No contraindication for adjuvant SoC endocrine treatment
15. No contraindication for elacestrant treatment
16. No contraindication for ribociclib treatment, if medically indicated, and adequate washout time for CYP3A4 inducers/inhibitors and QT time-prolonging drugs is given
17. Tumour block for central pathology review (core biopsy of initial diagnosis and biopsy/surgery sample of definite surgery), if available
18. Performance Status ECOG ≤ 1 or Karnofsky Index ≥ 80%
19. Laboratory requirements (female and male patients, not older than 14 days prior to date of informed consent)

    * absolute neutrophil count ≥ 1.5 × 109/L,
    * platelets ≥ 100 × 109/L,
    * haemoglobin ≥ 9.0 g/dL,
    * INR ≤ 1.5,
    * serum creatinine < 1.5 × ULN OR clearance ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
    * total bilirubin < ULN, except for patients with Gilbert's Syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN,
    * aspartate transaminase (AST) < 2.5 × ULN,
    * alanine transaminase (ALT) < 2.5 × ULN,
    * Screening lipid panel fasting levels: total cholesterol ≤400 mg/dL AND/OR triglycerides <500 mg/dL.

    Note: Patients with lipid panel fasting levels NOT meeting the above criteria may consider initiating therapy for lipid management per local guidelines and will be allowed to be included once the lipid levels meet the inclusion criteria.
20. Clinical assessments:

    • normal electrocardiogram within 6 weeks prior to randomization (QTcF interval at screening <450msec using Fridericia's correction, mean resting heart rate 50-90 bpm)
21. Ability to swallow tablets
22. Contraception

A. Female patients of childbearing potential at inclusion must have a negative pregnancy test (serum) and additionally fulfil either one of the following conditions:

* surgically sterile,
* or carry a non-hormone releasing intrauterine device (combined with a barrier method),
* or having received tubal ligation/occlusion (combined with a barrier method),
* or using a highly effective contraceptive method from the time they sign consent, during participation in the study until end of study, at least 4 months (120 days) after the last dose of ELA, and for at least 21 days after the last dose of RIBO) to prevent pregnancy; ova donation or preservation is also not allowed within this time frame
* Total/true abstinence: When the patient refrains from any form of sexual intercourse and this is in line with their usual and/or preferred lifestyle; this must continue from the time they sign consent, during participation in the study until end of study, at least 4 months (120 days) after the last dose of ELA, and for at least 21 days after the last dose of RIBO) to prevent pregnancy;
* Vasectomised sexual partner (with participant assurance that partner received post-vasectomy confirmation of azoospermia) combined with a barrier method or sexual partner with bilateral orchiectomy.
* Hormonal contraception is not acceptable. B. Male patients must either be
* surgically sterile
* or using a highly effective method of contraception from the time they sign consent, during participation in the study until end of study, at least 4 months (120 days) after the last dose of ELA, and for at least 21 days after the last dose of RIBO) to prevent pregnancy in a partner; sperm donation or preservation is also not allowed within this time frame
* Male patients who intend to be sexually active with a woman of childbearing potential, must use a condom plus spermicide from the time they sign consent, during participation in the study until end of study, at least 4 months (120 days) after the last dose of ELA, and for at least 21 days after the last dose of RIBO) to prevent pregnancy in a partner;
* Highly effective methods of contraception should be considered in female partners of men taking elacestrant and/or ribociclib who are of childbearing potential.

Exclusion Criteria:

1. Known hypersensitivity to any of the compounds or incorporated substances of the IMPs
2. Prior malignancy with a disease-free survival of <5 years, except curatively treated basalioma of the skin or pTis of the cervix uteri
3. Any history of invasive cancer within the last 10 years Note: adequately treated, basal or squamous-cell skin carcinoma, non-melanomatous skin cancer, curatively resected cervical cancer, and contralateral DCIS treated by mastectomy (contralateral in relation to current invasive breast cancer diagnosis) are excepted. Previous ipsilateral DCIS, irrespective of treatment, is excluded!
4. Patient with distant metastases of breast cancer beyond regional lymph nodes.
5. Concurrent treatment with cytotoxic agents for any non-oncological reason unless clarified with sponsor
6. Concurrent treatment with other experimental drugs
7. Participation in another interventional clinical trial with or without any investigational, not marketed drug within 30 days or 5 half-lives of the respective drug, whichever is longer, prior to study entry. In case of other interventional trial contact Sponsor.
8. Previous treatment (>4 weeks) with any SERD
9. Concurrent pregnancy; patients of childbearing potential or potentially childbearing partners of male patients must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
10. Breast feeding woman
11. Use of oral, transdermal, injected, or implanted hormonal methods of contraception as well as hormonal replacement therapy (oestrogen or progesterone).
12. Reasons indicating risk of poor compliance
13. Patient not able to consent
14. Patient has not recovered from clinical and laboratory acute toxicities related to prior anticancer therapies to NCI CTCAE version 5.0 Grade ≤ 1.
15. Severe and relevant co-morbidity that would interact with the application of endocrine treatment of any kind or the participation in the study
16. For patients planned for ribociclib treatment: Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality, including any of the following:

    * history of myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry,
    * documented cardiomyopathy,
    * left ventricular ejection fraction (LVEF) < 50 % as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO),
    * long QT syndrome, family history of idiopathic sudden death, congenital long QT syndrome, or any of the following:

      * risk factors for Torsades de Pointe (TdP, polymorphic ventricular tachycardia in patients with long QT syndrome) including uncorrected hypokalaemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/ symptomatic bradycardia,
      * concomitant medications with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug),
      * inability to determine the QTcF interval,
      * clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left-bundle branch block, high-grade AV block (e.g., bi-fascicular block, Mobitz type II, and 3rd-degree AV block),
      * systolic blood pressure (SBP) > 160 or < 90 mmHg.
17. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small-bowel resection).
18. Uncontrolled infection requiring i.v. antibiotics, antivirals, or antifungals
19. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection. Patients should be tested for HIV prior to randomization if required by local regulations or ethics committee (EC). Patients who test positive for HIV-antibody are excluded.
20. Patient has known active hepatitis-B-virus (HBV) or hepatitis-C-virus (HCV) infection. Screening for HBV or HBC-infection and testing for hepatitis-B or -C is highly recommended according to current valid (local) clinical guidelines, but neither part of the interventional study procedures, nor required for enrolment.
21. Patient has received live vaccines within 30 days prior to randomization.
22. Patient was submitted to an institution by virtue of an order of a court or a governmental authority must be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1520 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2033-09-30 (Estimated); Study Completion 2033-09-30 (Estimated)

PRIMARY OUTCOMES:
5-year invasive disease-free survival (iDFS) | iDFS 5 years
  iDFS after 5 years, compared between patients randomized to adjuvant elacestrant (+/-CDK4/6i) or SOC ET (+/- CDK4/6i)

SECONDARY OUTCOMES:
5-year distant disease-free survival (dDFS) | dDFS 5 years
  5-year dDFS
5-year relapse-free survival (RFS) | RFS 5 years
  5-year RFS
5-year DCIS disease-free survival (DFS-DCIS) | DFS-DCIS 5 years
  5-year DFS-DCIS
5-year invasive breast cancer-free survival (IBCFS) | IBCFS 5 years
  5-year IBCFS
5-year locoregional relapse-free survival (LRFS) | LRFS 5 years
  5-year LRFS
5-year overall survival (OS) | OS 5 years
  5-year OS

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schmid, PHD Dr, Principal Investigator — Fliethstraße 112-114 41061 Moenchengladbach Germany; NAdia Harbeck, Prof Dr, Principal Investigator — Breast Centre, Dept. Obstetrics & Gynaecology and CCC Munich LMU University Hospital Munich Germany; Oleg Gluz, Prof Dr, Principal Investigator — Breast Centre, Evang. Bethesda-Hospital Moenchengladbach Germany; Sherko Kuemmel, Prof Dr, Principal Investigator — Breast Centre, Kliniken Essen Mitte Essen Germany; Monika Graeser, PD Dr, Principal Investigator — Breast Centre, Marien-Hospital Witten Germany

IPD SHARING:
Plan to Share IPD: No